CLINICAL TRIAL: NCT01520662
Title: Impact of a Wellness Portal on The Delivery of Patient-Centered Preventive Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, James Mold, Professor, Director of Research Division, Agency for Healthcare Research and Quality (AHRQ)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Wellness Portal Study; 1R18HS017188-01 (AHRQ)
Record Dates: First submitted 2012-01-19; First posted 2012-01-30 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2012-01

CONDITIONS: Patient-centered Care
Keywords: patient-centered care; wellness; preventive services; primary care; To accomplish Aim 2, we will conduct a nine-month pre-post; randomized controlled trial (RCT) in four primary care; practices. The study will focus on the impact of a patient; Wellness Portal on the quantity and quality of preventive; care patients receive in primary care practices.

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wellness Portal Intervention (Experimental): Wellness Portal Intervention: patients have access to the portal in the course of the study.
  Interventions: Other: Implementation of a secure web-based patient Wellness Portal
- Wellness Portal Control (No Intervention): Control patients don't have access to the Wellness Portal in the course of the study.

INTERVENTIONS:
Other: Implementation of a secure web-based patient Wellness Portal — Patients in intervention practices will review and update their wellness records, risk factor information, allergy and contraindication profile, and personal preferences through the Wellness Portal before they visit their primary care provider.
  Arms: Wellness Portal Intervention

SUMMARY:
Building upon our experience with a very sophisticated preventive services prompt and reminder system, the Preventive Services Reminder System (PSRS), the investigators propose to conduct a systematic three-year study with the following aims:

1. To develop, field test, and refine an Internet-based patient Wellness Portal linked to PSRS to facilitate patient-centered, preventive care in primary care practices;
2. To determine the impact of the Wellness Portal on the process of patient-centered preventive care by examining the behavior and experiences of both patients and providers and the degree to which recommended services are individualized; and
3. To develop model Wellness Portal practices and disseminate the Wellness Portal technology and knowledge derived from Aims 1 and 2 findings.

DETAILED DESCRIPTION:
Project Aim 1: Develop, field test, and further refine an Internet-based Wellness Portal for use by patients seen in primary care settings to facilitate patient-centered, preventive care.

Specific Objectives:

* Assemble an Advisory Committee of clinicians, office staff, patients, and national HIT experts and develop a patient Wellness Portal that can be accessed by patients through the Internet and also in the provider's office via computer kiosks;
* Field test the Wellness Portal in two OKPRN practices and collect patient and provider satisfaction data via surveys and personal feedback to improve and refine the Wellness Portal and its integration into the comprehensive care delivery process.

Project Aim 2: Determine the impact of the Wellness Portal on the process of patient-centered preventive care by examining the experience of patients and providers with care and individualization of recommended services.

Specific Objectives:

* Assess the impact of the Wellness Portal on patient-centered care:

  1. Assess the impact of the Wellness Portal on patient activation and the medical home;
  2. Understand the impact of Wellness Portal use, the role of activated patients, and the concept of medical home on the provision of patient-centered care;
  3. Measure the impact of the Wellness Portal on the individualization of preventive services that are recommended and delivered based upon individual risk factors and patient preferences;
* Describe utilization and implementation of the Wellness Portal, capture and analyze documented decisions on opting out from evidence-based recommendations, and assess the impact of the portal on missed opportunities for delivering preventive care.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been seen at least twice by the enrolled clinician in the last twelve months;
* Patients must be six years old or younger or 50 years old and older;
* Patients (or their caretakers) must speak either English or Spanish and must have a basic level of computer skills that include being able to navigate a simple, consumer-oriented web site, use the keyboard and the mouse to interact with the browser, and understand / respond to

Exclusion Criteria:

* Not established patient
* Between than 6 years old and 50 years old
* Not fluent in English or Spanish, no basic computer skills or no help available for navigating a web browser

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2007-09; Primary Completion 2008-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Determine the impact of the Wellness Portal on the process of patient-centered preventive care by examining the experience of patients and providers with care and individualization of recommended services | 9 months run per practice / 12 months total

SECONDARY OUTCOMES:
a) Assess the impact of the Wellness Portal on patient-centered care b) Describe utilization and implementation of the Wellness Portal | 09/01/2007 - 08/31/2010

CONTACTS AND LOCATIONS:
Overall Officials: James W Mold, MD, MPH, Principal Investigator — University of Oklahoma HSC Department of Family and Preventive Medicine
Locations (1):
- University of Oklahoma HSC Department of Family and Prevetive Medicne, Oklahoma City, Oklahoma, United States

REFERENCES:
- See also: Home Page of the Oklahoma Physicians Resource/Research Network, a primary care practice-based PBRN — http://www.okprn.org